CLINICAL TRIAL: NCT05981534
Title: Double-blinded Randomized Controlled Trial Investigating the Effectiveness of Vitamin D Supplementation in Patients With End-stage Knee Osteoarthritis
Brief Title: The Effectiveness of Vitamin D Supplementation in Patients With End-stage Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.252
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Vitamin D Deficiency; Sarcopenia; Knee Osteoarthritis
Keywords: Vitamin D; Sarcopenia; Muscle atrophy; Knee Osteoarthritis
MeSH Terms: conditions — Vitamin D Deficiency; Sarcopenia; Osteoarthritis, Knee; Muscular Atrophy | interventions — Vitamin D; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive vitamin D supplement for 6 months
  Interventions: Drug: Vitamin D
- Control group (Placebo Comparator): The control group will receive placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 4000IU/day vitamin D supplement will be used for 6 months
  Other Names: SODX Co., Ltd, Osaka, Japan
  Arms: Intervention group
Drug: Placebo — Placebo will be used for 6 months
  Other Names: SODX Co., Ltd, Osaka, Japan
  Arms: Control group

SUMMARY:
Osteoarthritis (OA) knee is one of the commonest chronic degenerative conditions. It causes disability in elderlies due to pain and stiffness. The prevalence of radiologic knee osteoarthritis increases in proportion to age, reaching an astounding 64.1% for patients who are over 60 years of age. In 2021, there were over 26,000 patients on the Hospital Authority (HA) waiting list for knee total knee replacement (TKR) and with only 4300 TKRs performed, the nominal waiting time for TKR was almost 89 months.

Low vitamin D can adversely affect cartilage thickness and study suggested that low serum vitamin D is associated with increased radiographic knee OA progression. A systematic review concluded that vitamin D supplements can improve pain and function in patients with knee OA.

Vitamin D has long been recognized for its effect on musculoskeletal health and increasing attention has been focused for its effect on muscle function. Vitamin D have a direct effect on muscle hypertrophy by acting on specific vitamin D receptors (VDRs) on myocytes, and sufficient levels of vitamin D in patients have been found to correlate with an increase in the size, number, and strength of muscle fibres. Vitamin D also seems to exert beneﬁcial eﬀects by its interplay with myokines such as myostatin and irisin.

One study also showed that muscle nuclear VDR was increased by 30% and augmented muscle fibre size by 10% in elderly females (mean age of 78 years) taking vitamin D orally at a rate of 100 µg/day (4000 IU/day) for 4 months.

This will be a double-blinded RCT investigating the effect of vitamin D supplements or knee muscle strength, physical function, pain symptoms and, sarcopenia status. The study will be a follow-up study with assessment at baseline, 3- ,6-and 12-months post vitamin D intervention.

DETAILED DESCRIPTION:
Osteoarthritis (OA) knee is one of the common chronic degenerative conditions. It causes disability in elders, leading to pain and stiffness. The prevalence of radiologic knee osteoarthritis and symptomatic knee OA were 37.4% and 12.1% among adults over 60 years of age.

Often, patients with end-stage knee OA often adopt a sedentary lifestyle to avoid joint pain and stiffness. This can have an adverse effect on muscle function both locally around the knees as well as on generalized muscle health. Ageing and inactivity leads to a progressive loss of muscle mass and strength until an abnormally low level, termed "sarcopenia". Sarcopenic elderlies are more likely to develop deterioration of functional outcomes and higher mortality resulting in socioeconomic and healthcare burdens. In contrast, our previous study investigating the prevalence of sarcopenia in end-stage OA showed that 32.8% of severe knee OA patients also suffered sarcopenia, and these patients showed a slower recovery after undergoing TKR.

Vitamin D has long been recognized for its effect on musculoskeletal health, and increasing attention has been focused on its effect on muscle function. Vitamin D directly affects muscle hypertrophy by acting on specific vitamin D receptors (VDRs) in myocytes, and sufficient vitamin D levels in patients have been found to correlate with an increase in the size, number, and strength of muscle fibers. In the Chinese population aged over 65, 30.6% of the population studied presented with vitamin D deficiency (25(OH)D <20 ng/mL). A systematic review concluded that vitamin D supplements can improve pain and function in patients with knee OA. Moreover, patients with end stage OA knees will have more pain, leading to decreased mobility, a higher risk of sarcopenia, and vitamin D insufficiency that would warrant attention.

56 patients with end-stage knee OA scheduled for TKR will be recruited from the Li Ka Shing Orthopaedic Specialist clinic at the Prince of Wales Hospital (PWH) Hong Kong.

Oral and written consents will be obtained from individuals who agree to participate in the study.

The recruitment period will last for 12 months and the whole project period is 2 years in total. Basic demographics, sarcopenia assessment and Outcome Measurement Questionnaires will be carried out. The patients will be advised to avoid taking supplements and keep a record of medication intake throughout the study period.

We will use 4000 IU/day, for 6 months adapted from previous study. All study tablets including the placebo will be manufactured according to Good Manufacturing Practice (GMP) guidelines for quality assurance.

Assessments including quadriceps and hamstring muscle strength, handgrip strength, 6-meter timed walking gait test, chair stand test, muscle mass using Dual Energy X-ray Absorptiometry and questionnaires will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 50 with end-stage knee OA
* Patient are on the waiting list for TKR at Prince of Wales Hospital
* Walk unaided for 6 meters
* Able to comply with the assessments and has given oral and written consent
* Patients with vitamin D insufficiency and deficiency at the baseline measurement (25(OH)D <30 ng/mL)

Exclusion Criteria:

* Patients with connective tissue disorders or myositis condition
* History of any Hip & Knee surgery
* Patients with malnutrition were assessed by Mini-Nutritional assessment.
* Patients with acute immobility (i.e., post-hip fracture or post-acute hospital admission)
* Patient scheduled for TKR within six months
* Patients already taking vitamin D supplements
* Patients with a known contraindication to vitamin D treatment (such as allergy)
* Patients who have renal impairment with glomerular filtration rate (eGFR) < 30 ml/minute

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps and hamstring muscle strength assessment | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  Hand-held dynamometer microFET2 (Hoggan Scientific, Salt Lake City UT, USA) will be used to assess lower limb strength and power. Assessment of isometric muscle strength and power will be performed with the participants in a seated position to assess knee extensors and knee flexors. All tests will involve maximal voluntary isometric contractions. Both limbs will be assessed to record side-to-side difference. Two trials were recorded for each muscle group.

SECONDARY OUTCOMES:
The 6-meter timed walking test | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  The 6-meter timed walking test is a well-established test to assess gait speed. However, due to space limitations and the exhaustive nature of the test for patients with OA, the 6-meter test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
5-time Chair stand test | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  The chair stand test is a reliable test for assessment for low limb strength in patients. Patients will be asked to sit on a solid chair with arms on shoulders and feet with shoulder width apart. They will be instructed to do 1-2 repetitions to become familiar with the test, and perform as many reputations as they can in 30 seconds.
Dual Energy X-ray Absorptiometry (DXA) | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  The radiation for one session (20 minutes) for sarcopenia assessment is less than 25µSv, which is within the safe range. After every DXA scan, two copies will be printed that show the patients' body composition, bone mineral density, fat percentage, body mass index, and most importantly for this study, lean muscle mass.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  It is a questionnaire that measures a patient's pain, stiffness and physical function and can be summed up into a score out of 96. A high score indicates a more disabled participant .
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  To to evaluate symptoms and function in patients with knee injury and osteoarthritis with five separately scored subscales. Higher scores means better knee function
Short-Form 36 (SF-36) | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  36 questions to measure a patient's functional health and well-being from a patient's point of view. It is a reliable and validated measure that summarises the patients' physical and mental health. Higher scores means better quality of life.
International Physical Activity Questionnaire (IPAQ) | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  Assesses and monitors a patient's physical activity and inactivity level. This instrument sums up a patient's activity level per week into three categories, Category 1 Inactivity, category 2 minimally active and category 3 HEPA active
Nutritional intake questionnaire | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  Evaluation of habitual dietary intake will be based on retrospective means of assessment for the past twelve months. A Food Frequency Questionnaire (FFQ) previously validated with data obtained in the Hong Kong Adult Dietary Survey in 1995 as described previously will be used(Appendix 7). Daily dietary intake of Vitamin D and calcium will be evaluated by the Food Processor Nutrition Analysis and Fitness software version 7.9 (Esha Research, Salem, USA), with incorporation of local food composition based on food composition table from China
Sunlight exposure questionnaire | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  The Chinese version of the sunlight exposure questionnaire will be used in this study and has proven to be adequate for measurement of lifetime sunlight exposure among Hong Kong Chinese women. Higher scores means high chance of level vitamin D level.
Handgrip strength | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  The handgrip dynamometer will be used to test for the patients' handgrip strength. The handgrip dynamometer is an instrument measuring patients' maximum isometric strength of the hand and forearm muscles. The handle of the dynamometer will be adjusted as the finger is at 90 o whilst the dynamometer is being held. The measurement will be repeated three times and the average calculated for the dominant hand (Hand dominance will be determined by observing the patient's writing hand when signing the informed consent).
Serum myokine evaluation | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  Blood taking (5 ml) will be performed. The serum will be prepared by centrifugation and kept in a -80º freezer until use. Quantitative analysis for myokines and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities) or enzyme-linked immunosorbent assay (ELISA).
Serum vitamin D assays | Baseline, 3 months, 6 months, 12 months after the the commencement of vitamin D supplement
  Serum 25(OH)Vit-D levels will be measured by a commercial 25(OH) Vitamin D ELISA kit (Abcam ab213966) according to the manufacturer's instruction, providing the quantitative determination of 25(OH) Vitamin D3 and 25(OH) Vitamin D2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun ONG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewer

REFERENCES:
- [Derived] Wang QW, Ong MT, Man GC, Yeung YM, He X, Choi BC, Ng JP, Mok DK, Lam TP, Yung PS. The effectiveness of vitamin D supplementation in patients with end-stage knee osteoarthritis: Study protocol for a double-blinded, randomized controlled trial. PLoS One. 2024 Oct 21;19(10):e0309610. doi: 10.1371/journal.pone.0309610. eCollection 2024. PMID 39432457